CLINICAL TRIAL: NCT03824756
Title: Assessing the Effectiveness of Strengthening the Growth Monitoring and Promotional Activities in Improving the Nutritional Status of Children Under 2 Years of Age in Rural Bangladesh
Brief Title: Assessing the Effectiveness of Strengthening the Growth Monitoring and Promotional Activities in Rural Bangladesh
Acronym: GMP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PR-17123
Record Dates: First submitted 2019-01-17; First posted 2019-01-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-02

CONDITIONS: Nutritional Status
Keywords: Growth monitoring and promotion; child growth; Infant and young child feeding practices; program; Bangladesh

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NGO supported GMP program (Experimental): Intervention: NGO supported GMP program Site: Community clinic Duration: 12 months Study participants: 6-12 months aged children living within community clinic catchment area
  Interventions: Other: NGO supported GMP program
- Non-supported GMP program (Active Comparator): Comparison: Non-supported GMP program Site: Community clinic Duration: 12 months Study participants: 6-12 months aged children living within community clinic catchment area
  Interventions: Other: Non-supported GMP program

INTERVENTIONS:
Other: NGO supported GMP program — An International NGO has signed a contract with Government to support in implementing the growth Monitoring and Promotion (GMP) program. This program will be implemented at Community clinics. It will ensure the sustainability of community clinics in the selected areas through capacity building and follow up with community groups, community support groups, and Government Health and Family Planning service providers.
  Other Names: Intervention arm
  Arms: NGO supported GMP program
Other: Non-supported GMP program — This is control arm of the study. In this arm, there will be Government's usual GMP program implemented at community clinics without any NGO support.
  Other Names: Control arm
  Arms: Non-supported GMP program

SUMMARY:
Background: To tackle the high burden of undernutrition, the government of Bangladesh has identified growth monitoring and promotion (GMP) as a priority activity in the National Nutrition Services operational plan. Till date, no evidence are available from Bangladeshi studies to identify the effectiveness of GMP in improving the nutritional status of Bangladeshi children under 2 years of age. During 2013-14, two Bangladeshi studies looking at implementation issues of GMP at Community Clinic level and assessing the quality of nutrition services at primary health care facilities. The studies identified that lack of coordination, inadequate training, supervision, and logistic supplies as challenges to GMP implementation. Currently, GMP, (primarily sick child GMP) is being implemented through community clinics, supported by non-governmental organizations (NGOs) or other programs funded by donors. Besides, GMP is also taking place in areas where there are no NGO or donor support activities. However, the quality of nutrition data related to GMP is believed to be unsatisfactory. Hence, it is important to assess the effectiveness of GMP on the growth of under 2-year-old children.

Hypothesis: GMP services could improve the growth of children under 2 years of age by 20 percent in the intervention group compared to the control group

Objectives:To examine the effectiveness of GMP in improving nutritional status of children under 2 years of age

Methods:

Study design: Quasi-experimental study using mixed methods Study duration: 24 months Study setting: The study will be conducted in six sub-districts of rural Bangladesh where GMP is operational at the community clinic level. However, those areas will be excluded if there is any ongoing community or household level intervention on nutrition counseling being implemented by an NGO. For smooth implementation of GMP, refresher training on nutrition to health service providers will be provided by the study team.

Study participants: children under 2 years of age, mother's/caregiver's of children <2 and service providers.

Intervention group: children under 2 years of age who are exposed to GMP services at community clinics where an NGO funded program is supporting GMP implementation Control group: children under 2 years of age, at community clinics where GMP is not operational

DETAILED DESCRIPTION:
Introduction and objective:

Bangladesh has partly achieved the millennium development goal targets for nutrition and is committed to achieving the Sustainable development goals targets. Between 1997 and 2014, childhood stunting reduced from 60% to 36% nationally, and wasting has declined from 21% to 14%. However, 6.4 million children remain stunted, leaving them unable to develop to their full physical and mental potential. To tackle the high burden of under-nutrition, the government of Bangladesh has identified growth monitoring and promotion (GMP) as a priority activity in the National Nutrition Services operational plan. GMP is to be implemented from all primary health care facilities of the government health system. Growth Monitoring and Promotion (GMP) is a preventive activity comprised of growth monitoring linked with promotion (usually counseling) that increases awareness about child growth and improves caring practices. Ideally, in GMP, the weight of children usually under 2 years of age is measured periodically (for example, on a monthly or bi-monthly basis). The measurement can start at birth, accurately recorded on a growth chart, interpreted and explained to the caregivers. Additionally, the health workers give information through counseling, facilitating communication, and interacting with mothers in a way that aims to generate adequate maternal action to promote child growth. Recent systematic reviews question the effectiveness and relevance of GMP programs in general. Currently, GMP, which is primarily focused on sick child GMP is being implemented through community clinics (CCs), supported by NGOs or other programs funded by donors. Besides, GMP is also taking place in areas where there are no non-governmental organization (NGO) or donor support activities. However, the quality of nutrition data related to GMP is believed to be unsatisfactory. On this backdrop, it is important to assess the GMP implementation and its effect on the growth of under 2-year-old children. Hence, this study will offer a useful opportunity to examine the effectiveness of strengthening the GMP activities in improving growth and infant and young child feeding (IYCF) practices among children under 2 years of age in rural Bangladesh.

Selection of study site:

From the discussion and list of sub-districts shared by the NGO program, the investigators have selected 3 sub-districts where the program will be implemented from January 2018. The investigators have selected these 3 sub-districts based on (a) time of implementation of the program which matches with the project timeline; (b) available staff and logistics support by the NGO program in these sub-districts; and (c) large number of Community Clinics in these sub-districts to satisfy the required number of study participants and their caregivers. Additionally, the investigators have also selected 3 sub-districts as control keeping an adequate buffer zone to avoid intervention spill-over effect. The investigators will select 30 community clinics from these sub-districts through a community scoring system to have the maximum impact of the program.

Selection of study participants: The community clinics (CCs) and its catchment area will be considered as clusters. From the list of community clinics, required numbers of clusters will be randomly selected through a proportionate sampling. From the randomly selected CCs, the required number of study participants will be enrolled after conducting household listing.

Data collection procedures: The children will be enrolled from the catchment area of community clinics and be followed up for 12 months. During the follow-up period, the children will be visited periodically to assess their exposure to GMP service and also their feeding practice. Anthropometric measurements will be taken at baseline and then tri-monthly till the end of the 12 months follow-up period. Mother's knowledge and attitude about IYCF issues will be assessed at baseline and at an endpoint survey. Service provider's skills and perception about GMP will be assessed at baseline and at end-line. Quality of GMP implementation will be at baseline and periodically during the follow-up period.

Data collection tools: Household surveys, key informant interviews (KII), and observation.

Data analysis The survey data will be analyzed using STATA software (version 13). The summary statistics would be expressed as means with standard deviations, medians or percentages, with 95% confidence intervals (CI) where appropriate. To assess differences in mean among the factories, ANOVA and for categorical outcomes, chi-square statistical comparisons of proportions with 95% confidence intervals, will be calculated. A difference-of-difference (DID) analysis of quantitative outcome data will be done. To identify significant predictors associated with the main outcome indicators, bi-variate and multiple regression analyses will be employed.

Thematic analysis will be followed for qualitative information collected through participant's caregiver interview, key informant interview, and observation. Following preparation of the transcript, responses will be coded according to themes (a priori), sub-themes and emergent issues, if any. Triangulation of data derived from different methods will be carried out to validate qualitative information.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged between 6-12 months living in community clinic catchment area
2. Free from any acute or chronic illness(es)
3. Not a known case of a congenital anomaly or chromosomal abnormality
4. Not severely stunted (length-for-age Z score, LAZ <-3) or wasted (weight-for-length Z score, WLZ <-3) or underweight (weight-for-age Z score, WAZ <-3)
5. Not enrolled in any other intervention program
6. Caregiver report to have no plans to move out of the catchment area for at least 6 months following enrolment in the study

Exclusion Criteria:

Children's parents who will decline consent will not be enrolled in the study

-

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2000 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in length of the children under 2 years of age | 12 months
  Children who are aged between 6-12 months, their length in centimeter will be measured at baseline and then 3 monthly till end-line using a standard length board. The length for age z-score will be calculated by using a software developed by World Health Organization. The changes in length for age z-score will be detected through comparing the measurements over time by using difference-in-difference method.
Change in weight of the children under 2 years of age | 12 months
  Children who are aged between 6-12 months, their weight in kilograms will be measured at baseline and then 3 monthly till end-line using a standard weighing scale. The weight for age z-score will be calculated by using a software developed by World Health Organization. The changes in weight for age z-score will be detected through comparing the measurements over time by using difference-in-difference method.

SECONDARY OUTCOMES:
Change in mother's knowledge and attitude on infant and young child feeding (IYCF) practices measured by a standard semi-structured questionnaire | 12 months
  The change in IYCF practice will be reported in percentages through baseline and end-line differences through following indicators (either combined or separately):
  1. Early initiation of breastfeeding
  2. Introduction of solid, semi-solid or soft foods
  3. Minimum dietary diversity
  4. Minimum meal frequency
  5. Minimum acceptable diet: It summed the results of Minimum dietary diversity and Minimum meal frequency.
Changes in service provider's skill and perception on GMP | 12 months
  The community clinic service provider's skill and perception on GMP will be measured by using observation checklist and key informant interviews at baseline and end-line. The responses gathered from this 2 time points will be compared at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Muttaquina Hossain, MPH, Principal Investigator — Assistant Scientist

IPD SHARING:
Plan to Share IPD: No
The privacy, anonymity, and confidentiality of data/information identifying the study participants will be strictly maintained. Personal identifications taken during the survey will be kept under lock and key. None other than the study personnel will have access to information on personal identification and other sensitive information.

REFERENCES:
- [Derived] Hossain M, Ferdous TE, Islam Z, Billah SM, Bulbul MMI, Rahman MM, Ahmed T. Protocol for a quasiexperimental study testing the effectiveness of strengthening growth monitoring and promotion in community clinics for improving the nutritional status of under-two children in rural Bangladesh. BMJ Open. 2019 Oct 10;9(10):e032458. doi: 10.1136/bmjopen-2019-032458. PMID 31601604